CLINICAL TRIAL: NCT05277844
Title: A Phase II Randomized Controlled Trial of TKI Alone Versus TKI and Local Consolidative Radiation Therapy in Oncogene Driver Mutated Oligo Metastatic Non Small Cell Lung Cancer Patients
Brief Title: Local Consolidative Radiation Therapy Plus TKI Versus TKI Alone in Driver Mutated OM-NSCLC
Acronym: TARGET-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Anil Tibdewal, Principal investigator, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3338; CTRI/2019/11/021872 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2022-02-22; First posted 2022-03-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Oligometastatic Disease; Non-small Cell Lung Cancer; Driver Mutation
Keywords: Oligometastatic NSCLC; Driver mutation; TKI; Local consolidative therapy; SABR; Oligometastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Open-label, parallel-group RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Continuation of TKI therapy alone (Active Comparator): Patients in this arm will continue to receive standard treatment of TKI alone
  Interventions: Drug: TKI
- Arm 2: Continuation of TKI therapy + Local Consolidative Radiation therapy to 1-5 sites (Experimental): Patients will receive local consolidate radiation therapy to all oligo-metastatic sites plus radiation therapy to primary disease in addition to TKI
  Interventions: Radiation: Local Consolidative Radiation Therapy; Drug: TKI

INTERVENTIONS:
Radiation: Local Consolidative Radiation Therapy — Local consolidative radiation therapy to loco-regional disease and all Oligometastatic sites in addition to TKI
  Arms: Arm 2: Continuation of TKI therapy + Local Consolidative Radiation therapy to 1-5 sites
Drug: TKI — TKI

SUMMARY:
A Phase II randomized controlled trial of TKI Alone versus TKI and Local Consolidative Radiation Therapy in oncogene driver mutated oligo metastatic Non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Randomization Arms: Eligible patients will be randomized in 1:1 ratio to TKI alone or TKI + LCRT. This will be an intention to treat randomized study.

Arm 1: Continuation of TKI therapy alone Arm 2: Continuation of TKI therapy + Local Consolidative Radiation therapy to loc0-regional disease and 1-5 oligometastatic sites

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically proven diagnosis of NSCLC
2. Patients with positive oncogene driver mutation (EGFR or ALK/ROS)
3. Patients who have received at least 2-4 months of TKI therapy without progression
4. Patients with 1-5 sites of metastatic disease not including the primary tumor and regional nodes (less than 3 metastatic lesions in one organ will be eligible and 4 or more metastatic lesions in one organ will be ineligible)
5. Patients suitable for local consolidative therapy
6. Adequate end-organ function CBC/differential obtained within 15 days prior to registration on study, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 500 cells/mm3;
   * Platelets ≥ 50,000 cells/mm3;
   * Hemoglobin ≥ 8.0 g/dl (Use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable);
7. Patients with ECOG performance status of 0-2
8. Age > 18 years
9. For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to study registration

Exclusion Criteria:

1. Patients with progressive disease after 2-3 months of initial TKI therapy
2. Patients with negative oncogene driver mutations (EGFR/ALK/ROS)
3. Patients not suitable for local consolidative radiation therapy
4. Patients who are not suitable for further continuation of TKI therapy due to toxicity
5. Severe, active co-morbidity defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * Transmural myocardial infarction within the last 6 months;
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
6. Patients with prior history of radiation therapy to thorax
7. Patients with second malignancy (Synchronous or Metachronous)
8. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Upto 2 years
  Progression Free Survival will be defined as the time from the date of randomization until the date of disease recurrence or progression is documented, or until death in the absence of recurrence, whichever is earlier.

SECONDARY OUTCOMES:
Overall survival (OS) | Upto 2 years
  Overall survival will be defined as the time from randomization until the date of death from any cause in the presence or absence of recurrence.
Local control rates | Upto 2 years
  Local control will be defined as the lack of progressive disease at the treated sites (complete response, partial response and stable disease).
Health Related Quality of Life using the EORTC-QLQ-C30 questionnaire | From time of randomization to time of death or up to 24 months
  Quality of life will be assessed for each arm
Health Related Quality of Life using the EORTC-LC13 questionnaire | From time of randomization to time of death or up to 24 months
  Quality of life will be assessed for each arm
Toxicities using CTC v5.0 (radiotherapy related) | From time of Randomization to time of death or up to 24 months
  Toxicity will be defined as per the common terminology criteria version 5.0 at baseline and at subsequent follow up till 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anil Tibdewal, MD, Principal Investigator — Tata Memorial Hospital, Parel, Mumbai, Maharashtra, India
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
Protocol manuscript is published and the results will be published in International peer-reviewed journal

REFERENCES:
- [Background] Tibdewal A, Agarwal J, Mummudi N, Noronha V, Prabhash K, Patil V, Purandare N, Janu A, Kaushal R, Kannan S. Protocol for a phase II randomised controlled trial of TKI alone versus TKI and local consolidative radiation therapy in patients with oncogene driver-mutated oligometastatic non-small cell lung cancer. BMJ Open. 2021 Feb 15;11(2):e041345. doi: 10.1136/bmjopen-2020-041345. PMID 33589450